CLINICAL TRIAL: NCT02987881
Title: Physical Activity and Nutrition Counseling Intervention in Endometrial Cancer Survivors
Brief Title: Endometrial Cancer Diet and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Duke Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00074542
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2019-06

CONDITIONS: Early Stage Endometrial Cancer
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult women with early stage localized endometrial cancer (Experimental): Adult women with early stage localized endometrial cancer at least 2 months following hysterectomy
  Interventions: Behavioral: Home-based aerobic exercise and nutritional counseling

INTERVENTIONS:
Behavioral: Home-based aerobic exercise and nutritional counseling — Moderate walking and running with nutritional counseling at study visits.

SUMMARY:
This study will evaluate whether the use of the Jawbone wristband monitor, in connection with home-based exercise and nutritional counseling can be safely completed and improve cardiorespiratory fitness (heart and lung health) in women with early stage endometrial cancer who have undergone surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ages > 18 years.
* Localized endometrial cancer (stage I and II); no evidence of stage III or IV disease.
* At least 2 months was passed since the hysterectomy and enrollment.
* Karnofsky performance status > 70%.
* Body mass index of 30.0 - 49.9 and body weight < 300 pounds.
* No plan for adjuvant endometrial cancer therapy.
* Able to exercise safely on a treadmill.
* No absolute contraindications to exercise testing as recommended by the American Thoracic Society. No recent (<6 months) acute cardiac event unstable angina, uncontrolled dysrhythmias causing symptoms or hemodynamic compromise, symptomatic aortic stenosis, uncontrolled symptomatic heart failure, acute pulmonary embolus, acute myocarditis or pericarditis, suspected or known dissecting aneurism and acute systemic infection.
* The subject is not participating in regular physical exercise (more than 60 minutes of moderate intensity or 30 minutes of vigorous intensity exercise per week) or weight reduction dieting.
* Able to provide informed consent.
* Have reliable transportation to the testing facilities.
* Subjects must be able to speak and understand English to participate in this study.
* Subjects must have a personal mobile device compatible for the activity monitor

Compatible devices for the activity monitors are below:

* Android

  o Activity monitor is compatible with most Android devices equipped with Bluetooth 4.0 and running Android 4.3 (Jelly Bean) or later.
* iOS

  * iPhone 4s (or newer)
  * iPod touch (5th generation or newer)
  * iPad (3rd generation or newer)
  * iPad mini (1st generation or newer)
  * iPad Air (1st generation or newer)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by adherence to weekly walking sessions | Week 12
  Percentage of daily steps divided by total number of steps and daily walking sessions divided by total number of sessions prescribed
Safety as measured by the type and prevalence of adverse events during study-related assessments | Week 12
  Collection of events related to cardiopulmonary testing and self-reported events during off-site exercise training
change in cardiorespiratory fitness and CVD risk profile as measured by VO2peak | baseline and 12 weeks
change in cardiorespiratory fitness and CVD risk profile as measured by blood pressure | baseline and 12 weeks
change in cardiorespiratory fitness and CVD risk profile as measured by lipid profile | baseline and 12 weeks
change in cardiorespiratory fitness and CVD risk profile as measured by C-reactive protein | baseline and 12 weeks
change in cardiorespiratory fitness and CVD risk profile as measured by body composition | baseline and 12 weeks

SECONDARY OUTCOMES:
patient experience with exercise and nutrition counseling as measured by telephone questionnaire | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Angeles A Secord, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schwartz AR, Bartlett DB, Johnson JL, Broadwater G, Channell M, Nolte KC, Wilkes PA, Huffman KM, Secord AA. A Pilot Study of Home-Based Exercise and Personalized Nutrition Counseling Intervention in Endometrial Cancer Survivors. Front Oncol. 2021 Jun 11;11:669961. doi: 10.3389/fonc.2021.669961. eCollection 2021. PMID 34178654